CLINICAL TRIAL: NCT00829244
Title: A Phase IV Prospective, Multicenter, Randomized, Open-label Trial to Assess the Efficacy and Safety of GONAL f® at a Dose Based on Subject Baseline Characteristics Determined According to the CONSORT Calculator Compared With a Standard Dose of GONAL f® 150 IU Per Day for Ovarian Stimulation in Women Undergoing Assisted Reproductive Technology (ART)
Brief Title: CONSORT Randomized Controlled Trial in Assisted Reproductive Technology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28613
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Infertility
Keywords: Infertility; Assisted reproductive technology
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Glycoprotein Hormones, alpha Subunit

ARMS (2):
- CONSORT Dosing (Experimental): GONAL-f® dose based on subject baseline characteristics determined according to the CONSORT calculator
  Interventions: Drug: GONAL f® prefilled pen
- Standard Dosing (Active Comparator): GONAL-f® at a standard dose of 150 IU per day
  Interventions: Drug: GONAL f® prefilled pen

INTERVENTIONS:
Drug: GONAL f® prefilled pen — GONAL f® doses starting at minimum of 112.5 IU per day and a maximum of 450 IU per day for 1 cycle only
  Other Names: Follitropin alfa; Recombinant human follicle stimulating hormone (r-hFSH); GONAL-f® Prefilled Pen
  Arms: CONSORT Dosing
Drug: GONAL f® prefilled pen — GONAL f® standard treatment arm (150 IU of GONAL f® per day) up to Day 5 of stimulation after which the dose can be adjusted based upon the subject's ovarian response and according to the center's standard practice.
  Other Names: Follitropin alfa; r-hFSH; GONAL-f® Prefilled Pen
  Arms: Standard Dosing

SUMMARY:
The overall objective of this trial is to compare the ovarian response in assisted reproductive technology (ART) subjects administered GONAL f® according to the 'Consistency in recombinant follicle stimulating hormone [r-FSH] starting doses for individualized treatment' (CONSORT) calculator versus given a standard GONAL f® dose of 150 International Unit (IU) per day.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects justifying an in-vitro fertilization (IVF)/embryo transfer (ET) treatment
2. Have a male partner with semen analysis within the past 6 months prior to randomization considered adequate to proceed with regular insemination or intracytoplasmic sperm injection (ICSI) according to the center's standard practice. If these criteria are not met, the subject can only be entered if donor sperm will be used
3. Between her 18th and 35th birthday (35 not included) at the time of the randomization visit
4. Body mass index (BMI) lower than 30 kilogram per square meter (kg/m^2) where the BMI is calculated according to the formula
5. Have a regular spontaneous ovulatory menstrual cycle between 21 and 35 days in length
6. Have an early follicular phase (Day 2-4) serum level of basal FSH lower than or equal to 12 International Unit per Liter (IU/L) measured in the center's local laboratory during the screening period (i.e. within 2 months prior to down-regulation start)
7. Presence of both ovaries
8. Normal uterine cavity, which in the investigator's opinion is compatible with pregnancy
9. Have a negative cervical papanicolaou (PAP) test within the last 6 months prior to randomization
10. Have at least 1 wash-out cycle (defined as greater than or equal to 30 days since the last dose of clomiphene citrate or gonadotrophin treatment) since the last ART cycle and/or clomiphene citrate or gonadotrophin treatment prior to starting gonadotropin releasing hormone (GnRH) agonist therapy
11. Willing and able to comply with the protocol for the duration of the trial
12. Have given written informed consent, prior to any trial-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to her future medical care

Exclusion Criteria:

1. Have greater than or equal to 2 previous ART cycles with a poor response to gonadotrophin stimulation (defined as lower than or equal to 5 mature follicles and/or lower than or equal to 3 oocytes collected) or have greater than or equal to 2 previous ART cycles with a hyper response (defined as greater than or equal to 25 oocytes retrieved)
2. Any medical condition, which in the judgment of the investigator may interfere with the absorption, distribution, metabolism or excretion of the drug. In case of doubt, the subject in question should be discussed with Merck Serono's Medical responsible
3. Have previous severe ovarian hyperstimulation syndrome (OHSS)
4. Polycystic ovary syndrome (PCOS; Rotterdam criteria) to reduce the risk of the occurrence of OHSS
5. Presence of endometriosis requiring treatment
6. Uterine myoma requiring treatment
7. Any contraindication to being pregnant and/or carrying a pregnancy to term
8. Extra-uterine pregnancy within the last 3 months prior to screening
9. History of 3 or more miscarriages (early or late miscarriages) due to any cause
10. Tumors of the hypothalamus and pituitary gland
11. Ovarian enlargement or cyst of unknown etiology
12. Ovarian, uterine or mammary cancer
13. A clinically significant systemic disease
14. Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B or C virus in the trial subject or her male partner,
15. Abnormal gynecological bleeding of undetermined origin
16. Known allergy or hypersensitivity to human gonadotrophin preparations,
17. Any active substance abuse or history of drug medication or alcohol abuse in the past 5 years prior to the screening visit
18. Entered previously into this trial or simultaneous participation in another clinical trial

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Arriagada, MD, Study Director — Merck Serono S.A., Geneva
Locations (1):
- Research Site, Geneva, Switzerland

REFERENCES:
- [Derived] Olivennes F, Trew G, Borini A, Broekmans F, Arriagada P, Warne DW, Howles CM. Randomized, controlled, open-label, non-inferiority study of the CONSORT algorithm for individualized dosing of follitropin alfa. Reprod Biomed Online. 2015 Mar;30(3):248-57. doi: 10.1016/j.rbmo.2014.11.013. Epub 2014 Dec 15. PMID 25596910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 22 clinical trial centers in 9 European countries and 1 center in Chile. Recruitment period: 29 August 2008 to 21 January 2010.
Pre-assignment Details: A total of 244 participants gave informed consent and were screened for study entry. Forty-four (44) of these participants were not randomized due to: screening failure (38), failure to down regulate (3), or other reasons (3). A total of 200 participants were randomized to one of the two treatment arms.
Groups:
- GONAL-f ® CONSORT Calculator: GONAL-f® (follitropin alfa) administered subcutaneously (sc), dose ranging from 112.5 to 450 International Unit (IU) per day based on participant baseline characteristics determined according to the consistency in recombinant follicle stimulating hormone [r-FSH] starting doses for individualized treatment (CONSORT) calculator throughout stimulation cycle.
- GONAL-f ® Standard Treatment: GONAL-f® (follitropin alfa) administered sc at a standard dose of 150 IU per day up to Day 5 of stimulation (S5) after which the dose was adjusted based upon the participant's ovarian response and according to the center's standard practice.
Period: Overall Study
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Started | 96 | 104
Completed | 82 | 83
Not Completed | 14 | 21
Not completed — Adverse Event | 1 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of ovarian response to stimulation | 9 | 5
Not completed — Ovarian hyperstimulation syndrome (OHSS) | 1 | 6
Not completed — No fertilization | 2 | 2
Not completed — All embryos discarded | 0 | 3
Not completed — No embryo cleavage | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment | Total
Number analyzed (Participants) | 96 | 104 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 104 | 200
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Number of participants analyzed (N) = 86 and 93 for GONAL-f® CONSORT calculator and GONAL-f® standard treatment arm group respectively at screening.
  years | 30.0 (2.9) | 30.6 (2.6) | 30.3 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 104 | 200
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Chile | 7 | 8 | 15
  Denmark | 26 | 26 | 52
  France | 6 | 5 | 11
  Germany | 13 | 16 | 29
  Italy | 10 | 10 | 20
  Netherlands | 5 | 6 | 11
  Spain | 4 | 6 | 10
  Sweden | 8 | 7 | 15
  Switzerland | 11 | 14 | 25
  United Kingdom | 6 | 6 | 12
Serum Anti-Mullerian Hormone (AMH) [Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)] — Number of participants analyzed (N) = 86 and 93 for GONAL-f® CONSORT calculator and GONAL-f® standard treatment arm group respectively at screening.
  nanogram/milliliter (ng/mL) | 2.705 (1.870) | 2.399 (1.492) | 2.551 (1.692)
Serum Progesterone (P4) [Mean (Standard Deviation); unit: nanomole/liter (nmol/L)] — Number of participants analyzed (N) = 86 and 93 for GONAL-f® CONSORT calculator and GONAL-f® standard treatment arm group respectively at screening.
  nanomole/liter (nmol/L) | 2.934 (2.328) | 2.803 (2.291) | 2.868 (2.303)

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved Per Participant
Description: Mean number of oocytes retrieved on the day of ovum pick up (OPU) was calculated. Oocyte retrieval is a technique used in in-vitro fertilization in order to remove oocytes from the ovary of the female, enabling fertilization outside the body.
Time Frame: 34-38 hours post-recombinant human choriogonadotropin (hCG) (OPU)
Population: The modified Intention-To-Treat (ITT) population included all participants randomized into trial who received at least 1 dose of GONAL-f®, and who completed primary efficacy assessment (total number of oocytes retrieved per participant following GONAL-f® stimulation and hCG injection). Participants were analyzed based on treatment they received.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 86 | 93
oocytes | 10.0 (5.6) | 11.8 (5.3)
Statistical Analysis 1: Comparison: GONAL-f ® CONSORT Calculator vs GONAL-f ® Standard Treatment; The null hypothesis was that the difference between the mean number of oocytes [CONSORT calculator dosing - Standard dosing] was less than or equal to [=<] (-3). The alternate hypothesis was that the difference was greater than [>] (-3); Test type: Superiority or Other; p = 0.037, ANOVA; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-3.3 to -0.1], Standard Error of Mean 0.8

2. Secondary Outcome: Total GONAL-f® Dose
Time Frame: Start of treatment until end of stimulation cycle (approximately 28 days)
Population: The modified ITT population included all participants randomized into trial who received at least 1 dose of GONAL-f®, and who completed primary efficacy assessment (total number of oocytes retrieved per participant following GONAL-f® stimulation and hCG injection). Participants were analyzed based on treatment they received.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 86 | 93
IU | 1288.54 (300.95) | 1809.95 (546.90)
Statistical Analysis 1: Comparison: GONAL-f ® CONSORT Calculator vs GONAL-f ® Standard Treatment; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -511.37, 95% CI 2-sided [-638.78 to -383.96], Standard Error of Mean 64.52

3. Secondary Outcome: Mean GONAL-f® Daily Dose
Time Frame: Start of treatment until end of stimulation cycle (approximately 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 86 | 93
IU | 121.49 (22.56) | 167.43 (30.79)
Statistical Analysis 1: Comparison: GONAL-f ® CONSORT Calculator vs GONAL-f ® Standard Treatment; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Final Values) = -45.60, 95% CI 2-sided [-53.75 to -37.46], Standard Error of Mean 4.12

4. Secondary Outcome: Total Number of GONAL-f® Stimulation Treatment Days
Time Frame: Start of treatment until end of stimulation cycle (approximately 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 86 | 93
days | 10.6 (1.7) | 10.7 (1.6)
Statistical Analysis 1: Comparison: GONAL-f ® CONSORT Calculator vs GONAL-f ® Standard Treatment; Test type: Superiority or Other; p = 0.933, ANOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.5], Standard Error of Mean 0.2

5. Secondary Outcome: Number of Participants With Cancelled Cycles Due to Excessive or Inadequate Response to Treatment
Description: Number of participants with cancelled cycles due to excessive or inadequate response was evaluated. An excessive response: greater than or equal to 25 oocytes which could put the participant at risk of OHSS; An inadequate response: defined as 3 or less follicles of greater than or equal to 12 millimeter (mm) developing following at least 7 days of GONAL-f® treatment.
Time Frame: Start of treatment until Day 15-20 post-hCG
Population: All the randomized participants were analyzed for this outcome measure (N=200).
Measure: Number; unit: Participants
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 96 | 104
Participants
  Inadequate response | 9 | 5
  Excessive response (Risk of OHSS) | 1 | 6

6. Secondary Outcome: Percentage of Participants With Biochemical Pregnancies
Description: Biochemical pregnancy was defined as a pregnancy diagnosed only by the detection of hCG in serum and that does not develop into a clinical pregnancy.
Time Frame: Start of treatment until Day 15-20 Post-hCG
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 86 | 93
percentage of participants | 47.7 | 44.1
Statistical Analysis 1: Comparison: GONAL-f ® CONSORT Calculator vs GONAL-f ® Standard Treatment; Test type: Superiority or Other; Percent difference = 3.6, 95% CI 2-sided [-11.0 to 18.2]

7. Secondary Outcome: Number of Participants With Fetal Sacs and Fetal Hearts
Description: Number of participants with fetal sacs and fetal hearts (with activity) as seen on an ultrasound scan to confirm clinical pregnancy.
Time Frame: Day 35-42 Post-hCG
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 86 | 93
participants
  Missing (fetal sacs and fetal hearts) | 47 | 57
  0 (fetal sacs) | 6 | 1
  1 (fetal sacs) | 27 | 25
  2 (fetal sacs) | 5 | 10
  3 (fetal sacs) | 1 | 0
  0 (fetal hearts) | 8 | 3
  1 (fetal hearts) | 25 | 24
  2 (fetal hearts) | 5 | 9
  3 (fetal hearts) | 1 | 0

8. Secondary Outcome: Implantation Rate
Description: Implantation rate was measured as the number of gestational sacs observed divided by the number of embryos transferred multiplied by 100.
Time Frame: Day 35-42 Post-hCG
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent sacs per embryo
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 86 | 93
percent sacs per embryo | 31.1 (41.3) | 31.2 (40.8)
Statistical Analysis 1: Comparison: GONAL-f ® CONSORT Calculator vs GONAL-f ® Standard Treatment; Test type: Superiority or Other; p = 0.926, ANOVA; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-12.3 to 13.6], Standard Error of Mean 6.6

9. Secondary Outcome: Number of Participants With Multiple Pregnancies
Description: Multiple pregnancy was defined as 2 or more fetal hearts with activity.
Time Frame: Day 35-42 Post-hCG
Population: The modified ITT population. Number of participants analyzed (N) signifies those participants who were evaluated for this outcome measure.
Measure: Number; unit: participants
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 39 | 36
participants | 6 | 9

10. Secondary Outcome: Serum Progesterone (P4) Levels
Time Frame: End of stimulation cycle (approximately 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 86 | 93
nmol/L | 5.41 (7.57) | 4.88 (2.22)
Statistical Analysis 1: Comparison: GONAL-f ® CONSORT Calculator vs GONAL-f ® Standard Treatment; Test type: Superiority or Other; p = 0.235, ANOVA; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [-0.61 to 2.47], Standard Error of Mean 0.78

11. Secondary Outcome: Percentage of Participants With Clinical Pregnancy
Description: Clinical pregnancy is defined by the number of sacs and hearts with activity per ultrasound scan performed on Day 35-42 post-hCG.
Time Frame: Day 35-42 Post-hCG
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 86 | 93
percentage of participants | 36.0 | 35.5
Statistical Analysis 1: Comparison: GONAL-f ® CONSORT Calculator vs GONAL-f ® Standard Treatment; Test type: Superiority or Other; Percent difference = 0.6, 95% CI 2-sided [-13.5 to 14.6]

12. Secondary Outcome: Number of Participants With OHSS
Description: OHSS is a syndrome which can manifest with enlarged ovaries, advanced ascites with increased vascular permeability, pleural fluid accumulation, hemoconcentration, and increased blood clotting.
Time Frame: Start of treatment until Day 15-20 Post-hCG
Population: Safety population included all the participants who were randomized.
Measure: Number; unit: participants
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 96 | 104
participants | 6 | 13

13. Secondary Outcome: Pregnancy Outcome - Number of Participants With Pregnancy and Their Outcome
Description: Pregnancy outcomes are live outcome (live infant) and non-live outcome (non-live infant) or unknown outcome (subject lost to follow-up).
Time Frame: up to 9 month (following the end of treatment)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Number analyzed (Participants) | 31 | 33
participants
  Live outcomes | 24 | 25
  Non-live outcomes | 2 | 3
  Unknown outcomes | 5 | 5

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected on an ongoing basis from day of written informed consent. All new AEs must be recorded until the final treatment examination, on Day 15-20 of the post-treatment assessment period
Description: Pre-Treatment:Medical conditions present at the initial study visit that did not worsen in severity or frequency during the study; Treatment-Emergent: If the onset date of the AE was on or after the first dose date of the study medication.
Arm/Group | GONAL-f ® CONSORT Calculator | GONAL-f ® Standard Treatment
Serious Adverse Events (participants affected / at risk) | 4/96 | 3/104
Other Adverse Events (participants affected / at risk) | 40/96 | 48/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GONAL-f ® CONSORT Calculator (N=96) | GONAL-f ® Standard Treatment (N=104)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GONAL-f ® CONSORT Calculator (N=96) | GONAL-f ® Standard Treatment (N=104)
Nausea (Gastrointestinal disorders) | 8 (9) | 9 (11)
Abdominal distension (Gastrointestinal disorders) | 8 (8) | 3 (5)
Headache (Nervous system disorders) | 18 (30) | 25 (40)
Adnexa uteri pain (Reproductive system and breast disorders) | 9 (10) | 8 (9)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 5 (5) | 11 (12)
Procedural pain (Injury, poisoning and procedural complications) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall submit any results communication to the sponsor for review and comment at least 30 business days prior to submission. The sponsor shall have the right to request the PI to delete or modify any of sponsor's proprietary information contained therein. If the PI does not agree to the deletion or appropriate modification of such information, it shall postpone submission for publication or presentation for 60 days from the date the PI notifies the sponsor.